CLINICAL TRIAL: NCT06869395
Title: Alternative Therapies Prescribed by Pharmacists and Herbalists for Suspicious Oral Ulcer: a Cross-sectional Study
Brief Title: Alternative Therapies Prescribed by Pharmacists and Herbalists
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, PI, Cairo University
Other Study IDs: ACU-Med4
Record Dates: First submitted 2025-03-02; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prescription Drug Problems
Keywords: oral potentially malignant lesion
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — The responses obtained will be recorded as follows:
  - Referred to a dentist
  - Referred to a physician
  - Prescribed an over the counter (OTC) preparation
  - Prescribed an OTC preparation and referred to a dentist or a physician
  - Wanted to see the patient
  - Other answers: ………..

SUMMARY:
The cross-sectional study will recruit herbalists and pharmacists at their workplaces (herbal shops and pharmacies); where they will be asked their advice about a patient suffering from a potentially malignant condition.

DETAILED DESCRIPTION:
The cross-sectional study will recruit herbalists and pharmacists at their workplaces (herbal shops and pharmacies); where they will be asked their advice about a patient suffering from a potentially malignant condition.

Based on the standardized simulated patient approach, the cross-sectional study was planned in which an individual interacts with the interviewee according to a previously prepared script.

ELIGIBILITY:
Inclusion Criteria:

* working as herbalist, pharmacist or assistant pharmacist

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: herbalist, pharmacist or assistant pharmacist
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Referral to specialist | 2 months
  The pharmacists or herbalists are asked for their advice to the case: would they refer to specialist or not. It is a binary outcome (Yes/No)